CLINICAL TRIAL: NCT02091297
Title: Comparison of Transversus Abdominis Plane Block Versus Patient-controlled Epidural Analgesia for Patients on Buprenorphine or Methadone, After Cesarean Section
Brief Title: Comparison of Different Methods of Pain Control After Cesarean Section for Patients on Buprenorphine or Methadone
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: two other institutions that were in the center thought they weren't going to be able to recruit enough patients
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: D14074
Record Dates: First submitted 2014-03-10; First posted 2014-03-19 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Caesarean Delivery
Keywords: Buprenorphine; Suboxone; Subutex; Buprenex; Caesarean Delivery
MeSH Terms: interventions — Ropivacaine; Acetaminophen; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAP BLOCK (Active Comparator): One unique regional technique for lower abdominal surgery, that has been shown effective for Cesarean Section in particular, is the transversus abdominis plane (TAP) block, which blocks T6-L1 sensory nerve branches and provides anesthesia to the anterior abdominal wall. The TAP block has been recommended and shown in case reports, but not clinically studied with trials, for patients on methadone or buprenorphine, to improve post-operative pain control. A long active local anesthetic, called ropivacaine, will be used to provide this anesthesia.
  Interventions: Drug: TAP Block; Drug: Acetaminophen
- Common Care (Active Comparator): Common care refers to the common way pain is treated after Cesarean Section: a long-acting spinal or epidural opioid such as morphine, plus oral and IV opioids and non-narcotic adjuncts such as non-steroidal anti-inflammatory drugs and acetaminophen. Due to the potential issues such as ineffectiveness and fear of respiratory depression, increasing the dosing of these opioids may not be ideal.
  Interventions: Drug: Acetaminophen; Drug: Morphine
- Patient Controlled Epidural Analgesia (Active Comparator): For post-Cesarean analgesia, another regional technique that has been employed for superior pain control is continued epidural analgesia with local anesthesia and an opioid, either in addition or instead of long acting neuraxial opioids (Cohen). One study revealed equal analgesic efficiency, higher patient satisfaction scores, and less side effects with patient controlled epidural ropivacaine compared to epidural morphine (Chen). This is an especially attractive option for opioid dependent patients, but like the TAP block, has been not studied whether or not it lessens acute or chronic postoperative cesarean section, in the setting or in the absence of neuraxial opioids.
  Interventions: Drug: Ropivacaine; Drug: Acetaminophen

INTERVENTIONS:
Drug: TAP Block — This intervention of a TAP block will be compared to the intervention of Common Care and to the intervention of Patient Controlled Epidural Analgesia
  Arms: TAP BLOCK
Drug: Ropivacaine — The intervention of the Patient Controlled Epidural Analgesia will be compared to the intervention of a TAP block and the intervention of Common Care
  Arms: Patient Controlled Epidural Analgesia
Drug: Acetaminophen — Common ways to treat pain control after Cesarean Section include oral and IV opioids, non-narcotic adjuncts such as non-steroidal anti-inflammatory drugs and acetaminophen, and long-acting spinal or epidural opioids such as morphine. Due to the potential issues such as ineffectiveness and fear of respiratory depression, increasing the dosing of these opioids may not be ideal.
  The intervention of Common Care will be compared to the intervention of a TAP block and the intervention of Patient Controlled Epidural Analgesia
Drug: Morphine
  Arms: Common Care

SUMMARY:
More and more women are on buprenorphine or methadone during pregnancy for a history of opioid addiction. Currently, pain control after cesarean section for women already on these medications, if they need operative delivery, is a challenge due to the pharmacology of those drugs. They have higher pain scores and 45-47% higher opiates requirement. To improve pain control, some unique regional anesthesia techniques have been employed, besides opioid and non-opioid medication management through the oral, intravenous, and/or neuraxial (spinal or epidural) route. One is a TAP block ( transversus abdominis plane block), a regional anesthesia procedure in which long acting local anesthetic, such as ropivacaine, is injected on both sides of the patient's abdomen to numb the nerves supplying the abdominal wall, or the surgical site. Another is a patient - controlled epidural, a small flexible catheter that is inserted in the back into the epidural space near the spine, which bathes the spinal nerve roots with long acting local anesthetic, such as bupivacaine, and with an opioid, such as fentanyl, to numb the nerves going to the surgical site. Through an epidural pump, the patient receives a continuous infusion of local anesthetic and can delivery more medication as needed through a bolus feature. There have case reports, or case by case accounts, of these techniques, and it is suspected these techniques result in better pain control with minimal side effects. No clinical, human or animal, has evaluated these techniques in a controlled and through manner, either comparing the two techniques to each other or comparing them to the common care of opioid and non-opioid medication management through the oral, intravenous, and/or neuraxial route, including neuraxial hydromorphone or morphine.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiology Society of Anesthesiologist's Status of II or III
* Maintenance methadone or buprenorphine during pregnancy
* Regional anesthesia staff to perform a TAP block
* Elective, non-urgent cesarean delivery via a Pfannenstiel incision under regional anesthesia

Exclusion Criteria:

* Emergency cesarean section
* Laboring patients who are now having to delivery operatively
* Patients with a BMI over 50
* Patients with allergies to any of the study medications
* Patients under 18 years old
* Patients with multiple gestations
* Patients undergoing general anesthesia
* Patients who had contraindications for either an epidural or a TAP block as in coagulopathies, chronic back pain, skin conditions, or existing neuropathies
* Patients who cannot understand the use of a patient controlled epidural analgesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Acute pain by narcotic use after cesarean section | 0-48 hours after surgery
  Directly compare narcotic use in patients who have a TAP block, who have a patient - controlled epidural analgesia, or common care ( neuraxial opioid alone) while in the hospital / acute pain after Cesarean Section
  Will use morphine equivalents
Acute pain by pain scores after cesarean section | 0-48 hours
  Directly compare pain scores in patients who have a TAP block, who have a patient - controlled epidural analgesia, or common care ( neuraxial opioid alone) while in the hospital / acute pain after Cesarean Section
  Will use VAS (0-10), pain at rest, pain with movement

SECONDARY OUTCOMES:
Chronic pain by narcotic use | 6 weeks post-partum
  Directly compare narcotic use in the three groups at the six week visit, evaluating for chronic pain after Cesarean Section.
  Will use dose of buprenorphine and/or methadone Will use morphine equivalents
Respiratory depression | 0-48 hours
  Oxygen requirement, narcan use (yes / no), rapid response or code blue called
Perception of Quality in Anesthesia / Maternal Satisfaction | 0-48 hours
  Using the validated, "Perception of Quality in Anaesthesia (PQA) questionnaire", the patients assessed their overall experience of the cesarean section and post-operative pain management and anesthetic care
Pruritus | 0-48 hours
  Is a positive to pruritus if the patients answers yes to the question, "have you experienced any itching" or if a drug was specifically used to treat itching via a review of the MAR
Nausea | 0-48 hours
  Is a positive to nausea if the patients answers yes to the question, "have you experienced any nausea" or if a drug was specifically used to treat nausea via a review of the MAR
Vomiting | 0-48 hours
  Is a positive to vomiting if the patients answers yes to the question, "have you experienced any vomiting" or if a drug was specifically used to treat vomiting via a review of the MAR
Chronic pain by pain scores | 6 weeks post-partum
  Directly compare pain scores in the three groups at the six week visit, evaluating for chronic pain after Cesarean Section.
  Will use VAS score (0-10), pain at rest and pain with movement

CONTACTS AND LOCATIONS:
Overall Officials: Marnie B Welch, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Michaela Farber, MD, Study Director — Brigham and Women's Hospital; Lisa Leffert, MD, Study Director — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire